CLINICAL TRIAL: NCT06233773
Title: The Effect of Kinesio Taping and Manual Lymph Drainage on Syndrome Severity, Sleep Quality and Psychological Well-Being in Pregnant Women With Restless Leg Syndrome
Brief Title: The Effect of Kinesio Taping and Manual Lymph Drainage on Pregnant Women With Restless Legs Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: TC Erciyes University (Other)
Responsible Party: Principal Investigator, Ali Kaplan, Assist. Prof. Dr., TC Erciyes University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Supportive Care
Other Study IDs: Erciyes U - Ali KAPLAN
Record Dates: First submitted 2024-01-11; First posted 2024-01-31 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Pregnancy; Restless Leg Syndrome; Nursing
MeSH Terms: conditions — Restless Legs Syndrome | interventions — Manual Lymphatic Drainage; Control Groups

STUDY DESIGN:
Intervention Model Description: This research is a randomized controlled experimental study.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Kinesio Taping Group (Experimental): In this project, Kinesio Taping will be applied to the Kinesio Taping group to reduce pain and support circulation. In this study, space correction method to reduce pain and lymphatic correction technique to support circulation will be applied from Kinesio Taping methods. In the study, in order to determine the susceptibility to allergy to kinesio tape, a five cm application will be made on the outer lateral region of the arms of pregnant women and waited for 10 minutes. Before the application, the physiotherapist will clean the application area with volatile alcohol for correct and good adhesion of the tape. Four bands of 10 cm each will be cut for the application. In order to protect the tape during the movement of the person, all corners will be oval shaped and the kinesio tape will be adhered to the BL-40 and BL-57 points bilaterally using 25-50% tension with the space correction method.
  Interventions: Procedure: Kinesio Taping
- Manual Lymph Drainage Group (Experimental): Before the application, the pregnant woman will open both lower extremities, including the knee area, in a semi-sitting position. The other body parts will be covered with a sheet/sweater so that the leg area is open. Without applying anything (oil, vaseline, cream) to the leg, the physiotherapist will perform Manual Lymph Drainage using his/her hands. The pregnant woman will be asked to do 10 repetitions of diaphragmatic breathing exercise. Popliteal lymph nodes will be stimulated manually 7 times. The anterior and medial knee will be stimulated 7 times each with circular movements. Manual Lymph Drainage will be performed on the front of the leg with the pumping technique and on the back of the leg with the scooping movement. The procedure will be repeated 3 times to provide drainage in the same area. The ankle will be stimulated 7 times with circular movements. The inferior and posterior parts of both the medial malleolus and lateral malleolus will be stimulated.
  Interventions: Procedure: Manual Lymph Drainage
- Kinesio Taping and Manual Lymph Drainage Group (Experimental): In this group, Kinesio Taping and Manual Lymph Drainage will be performed together to support circulation and reduce pain. All of the procedures performed in the Kinesio Taping Group and the Manual Lymph Drainage Group will be performed in parallel. After Kinesio Taping, Manual Lymph Drainage will be performed for 6 days. The kinesio tape will be renewed on the fourth day and will remain for three more days.
  Interventions: Procedure: Kinesio Taping; Procedure: Manual Lymph Drainage
- Control Group (Active Comparator): Pregnant women in the control group will not be subjected to any intervention other than routine follow-up and care at the hospital.
  Interventions: Other: Control Group

INTERVENTIONS:
Procedure: Kinesio Taping — Kinesio Taping
  Arms: Kinesio Taping Group; Kinesio Taping and Manual Lymph Drainage Group
Procedure: Manual Lymph Drainage — Manual Lymph Drainage Group
  Arms: Kinesio Taping and Manual Lymph Drainage Group; Manual Lymph Drainage Group
Other: Control Group — Control Group
  Arms: Control Group

SUMMARY:
Restless Leg Syndrome, a progressive and recurrent chronic sensorimotor disorder that creates an irresistible urge to move the legs and a feeling of discomfort, is seen in 15.4-26.0% of pregnant women in our country. Restless Leg Syndrome has negative effects on sleep, mood, cognitive health, daily activities and behavior in pregnant women; It can also cause preeclampsia, difficult labor, and cesarean delivery. Therefore, it is important for pregnant women with Restless Leg Syndrome to be treated appropriately.

It is recommended that pregnant women use non-pharmacological treatments as they are not risky for fetal health. Kinesio taping and manual lymphatic drainage methods are used non-pharmacologically to support venous-lymphatic drainage and manage pain. These methods are economical, reliable and easy to apply. However, no study has been found in which Kinesio taping or manual lymphatic drainage was applied to a patient group with Restless Leg Syndrome during or outside pregnancy.

The aim of this project is to determine the effect of Kinesio taping and manual lymphatic drainage on Restless Legs Syndrome severity, sleep quality and psychological well-being in pregnant women with Restless Legs Syndrome.

DETAILED DESCRIPTION:
Restless Leg Syndrome, which creates an irresistible urge to move the legs, is seen in 15.4-26.0% of pregnant women in our country. Restless Leg Syndrome has negative effects on sleep, mood, cognitive health, daily activities and behavior in pregnant women; It can also cause preeclampsia, difficult labor, and cesarean delivery.

It is recommended that pregnant women use non-pharmacological treatments as they are not risky for fetal health. Studies have determined that progressive relaxation exercise and application of hot and cold water to the legs can reduce the severity of symptoms in pregnant women with Restless Leg Syndrome. However, the fact that progressive relaxation exercise covers a long period of time, such as eight weeks, may negatively affect the continuity of the practice in pregnant women. Due to the enlargement of the abdomen in the following weeks of pregnancy, pregnant women have difficulty in putting on and taking off compression stockings and sweat in the summer months; some pregnant women may experience negative effects when applying hot and cold water, such as heat sensitivity or the difficulty of repeating the application every evening. For this reason, it is necessary to increase the variety of non-pharmacological methods that can be recommended by healthcare personnel and by which pregnant women can choose the method most suitable for them in the symptom management of Restless Leg Syndrome that develops due to pregnancy. Kinesio taping and manual lymphatic drainage methods are used non-pharmacologically to support venous-lymphatic drainage and manage pain. These methods are economical, reliable and easy to apply. However, no study has been found in which Kinesio taping or manual lymphatic drainage was applied to the patient group with Restless Leg Syndrome during pregnancy or outside of pregnancy. Therefore, experimental studies evaluating the effectiveness of Kinesio taping and manual lymphatic drainage on Restless Leg Syndrome complaints are needed. This study will determine the effectiveness of Kinesio taping and manual lymphatic drainage in Restless Leg Syndrome complaints and provide evidence for the hypothesis that Restless Leg Syndrome may be associated with venous insufficiency. At the end of this project, if it is proven that Kinesio taping has an effect on complaints; a practical and ready-made Kinesio taping product development project that the pregnant woman can use on her own will be planned.

The aim of this project is to determine the effect of Kinesio taping and manual lymphatic drainage on Restless Leg Syndrome severity, sleep quality and psychological well-being in pregnant women with Restless Leg Syndrome. The study will be carried out at Erciyes University Hospital. Pregnant women who meet the inclusion criteria will be randomized into groups (Kinesio taping, manual lymphatic drainage, Kinesio taping + manual lymphatic drainage, Control), with 20 people in each group.

Data will be collected with Restless Leg Syndrome Diagnostic Criteria Survey Form, Research Criteria Compliance Form, Personal Information Form, Restless Leg Syndrome Severity Rating Scale, Richard-Campbell Sleep Scale, Psychological Well-Being Scale and Application Satisfaction Form.

After preliminary tests are performed, kinesio tape will be applied to Kinesio taping group's legs. Manual lymphatic drainage will be built for manual lymphatic drainage Group. Tape will be attached to Kinesio taping+manual lymphatic drainage group and manual lymphatic drainage will be made. No treatment will be applied to the control group. Tests will be repeated on the fourth and seventh days. SPSS program will be used to analyze the data.

Work packages of the study and by whom it will be carried out have been determined. Precautions and plans have been made for the risks that may develop in the project.

The experiences and knowledge gained at the end of the project will be shared by publishing articles or papers in international journals. In addition, it is expected that the scholars will increase their competencies in the field, develop a commercial product after the study, and create new studies or projects. Most importantly, a new method can be offered to pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age,
* Literate,
* Gestational week 13 and above,
* She has a singleton pregnancy,
* Presence of RLS according to the RLS Diagnostic Criteria Questionnaire and physician examination,
* A score of 11 or above on the RLS Severity Rating Scale,
* Pregnant women taking iron, vitamin D, magnesium and calcium will be included in the study.

Exclusion Criteria:

* Pre-pregnancy RLS,
* Communication barriers,
* Absolute bed rest for reasons such as cervical insufficiency, premature rupture of membranes or risk of preterm labor,
* Have any psychiatric illness, use antipsychotic and/or antidepressant medication,
* Acute infection of bacterial or viral origin,
* Varicose veins in the feet and legs and severe lymphedema (circumference difference between both extremities over 5 cm),
* Have a dermatologic problem in their feet and legs,
* Pregnant women with rheumatic diseases such as rheumatoid arthritis, osteoarthritis, ankylosing spondylitis, systemic lupus erythematosus, fibromyalgia will not be included in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Restless Leg Syndrome Diagnostic Criteria Survey Form | 13 months
  The diagnosis form was created by the International Restless Legs Syndrome Study Group in 1995, based on the patient's history. The form, with a Cronbach alpha coefficient of 0.81, consists of 5 questions. A diagnosis of Restless Leg Syndrome is made by answering "yes" to all questions on the form. The reliability and validity study of the form in Turkey was conducted.
Research Criteria Eligibility Form | 13 months
  The form created by the researchers will be used to determine whether pregnant women meet the eligibility criteria for the study. The form consists of two parts: inclusion criteria and exclusion criteria. Criteria are answered yes or no. In order for pregnant women to be included in the study, they must answer yes to all inclusion criteria and no to all exclusion criteria.
Personal Information Form | 13 months
  The form prepared by the researchers consists of questions containing socio-demographic and obstetric characteristics of women and a section containing lower extremity circumference measurement values of pregnant women.
Restless Leg Syndrome Severity Rating Scale | 13 months
  Scale was developed by the International Restless Legs Syndrome Study Group. The Restless Leg Syndrome Rating Scale, with a Cronbach alpha coefficient of 0.82, consists of 10 questions. Restless Leg Syndrome severity values in each question are graded as having no effect of Restless Leg Syndrome (0 points) or having a very severe effect (4 points). Thus, a total score is obtained, with the entire score range ranging between 0 and 40. The score between 1-10 indicates the presence of mild, the score between 11-20 indicates the presence of moderate, the score between 21-30 indicates the presence of severe, and the score between 31-40 indicates the presence of very severe Restless Leg Syndrome. A validity and reliability study of the scale was conducted in our country.
Richard-Campbell Sleep Scale | 13 months
  It was developed by Richards in 1987. The Richard-Campbell Sleep Scale consists of 6 items and this scale evaluates the depth of night sleep, the time it takes to fall asleep, the frequency of waking up, the time spent awake when waking up, the quality of sleep and the noise level in the environment. Each item of the scale is evaluated using the visual analog scale technique ranging from 0 to 100. A score of "0-25" from the scale indicates "very poor sleep" and a score of "76-100" indicates "very good sleep". When calculating the total score of the scale, the scores from 5 items are added together, and the 6th item, which evaluates the noise level in the environment, is not included in the total score evaluation. It is thought that as the scale score increases, the patient's sleep quality also increases.
Psychological Well-Being Scale | 13 months
  The scale was first named "Psychological Well-Being Scale", but its name was later revised to "Flourishing Scale", as it was thought that it would better express psychological well-being. The adaptation of the scale to Turkish was done, and the first name of the scale was used on the grounds that it was not the exact equivalent of the word flourishing. The scale, which consists of 8 items, is one-dimensional and contains positive expressions. The lowest score that can be obtained from the 7-point Likert type scale (between 1: Strongly disagree and 7: Strongly agree) is 8 and the highest score is 56. High scores on the unidimensional scale indicate a high level of psychological well-being. In the reliability study of the scale, the Cronbach's alpha internal consistency was calculated as 0.80 and the test-retest coefficient was calculated as 0.86, and it was stated that the scale is valid and reliable for use.
Application Satisfaction Form | 13 months
  The form was created by the researchers to determine the participants' satisfaction levels with the application. Satisfaction levels consist of two parts, where positive and negative feedback about the application is expressed numerically on a 10-point scale and open-ended. The form will be filled out by pregnant women at the end of the application along with the final test.

CONTACTS AND LOCATIONS:
Overall Officials: MÜRÜVVET BAŞER, Prof. Dr., Principal Investigator — Erciyes U
Locations (1):
- Erciyes University Medical faculty hospital, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No